CLINICAL TRIAL: NCT05416541
Title: Uncontrolled Disinformation About Regional Anesthesia From Social Media, and the Effect on the Pregnant Patients Decisions.
Brief Title: Uncontrolled Disinformation About Regional Anesthesia and Pregnant Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E1-21-1739
Record Dates: First submitted 2022-06-09; First posted 2022-06-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Regional Anesthesia; Anxiety; Social Media Addiction; Spinal Anesthesia; Fear Anxiety
Keywords: social media; anxiety; regional anesthesia
MeSH Terms: conditions — Anxiety Disorders; Internet Addiction Disorder | interventions — Media Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant patients
  Interventions: Behavioral: social media

INTERVENTIONS:
Behavioral: social media — ASA I-II, who speaks and writes Turkish and do not have psychiatric illness patients will attend the study.

SUMMARY:
Nowadays, hundreds of information about regional anesthesia are accessed from any internet search engine when a question is written about the methods of anesthesia that can be applied during C/S. This information may have positive or negative effects on the patient, as well as include uncontrolled, unsupervised comments, articles and images. Our aim is primarily to evaluate whether our patients are exchanging information via social media or the internet and the effects of these shares on their concerns.

DETAILED DESCRIPTION:
Social media has become a place to receive and share information today, especially for women of childbearing age. according to a study published in 2019, 78% of social media users are women and 80% of them are in the 18-40 age range. Again, studies have shown that women often use a large number of alternative platforms to receive or share information about pregnancy and parenting.

It has been shown that there are 3 different reasons why patients follow medical content on social media. Behaviorally, patients can be self-healing with the information they receive; cognitively, the search for information about their own condition and the desire to understand their condition is the desire to be able to share common feelings with other people who are in the same situation emotionally.

Anxiety develops in the preoperative period in 21-25% of cesarean section patients. This anxiety response can cause premature and low birth weight baby birth by vasoconstricting the uterine artery through the autonomic central nervous system.

It is common for pregnant women who already have concerns before the cesarean section that will take place to look for information about both the surgery and the anesthesia method that will be applied. Studies including patients who were watched preoperative anesthesia videos about the anesthesia technique, has showed low anxiety levels. However, this videos were custom made videos by the organizations such as hospitals, universities.

Nowadays, hundreds of information about regional anesthesia are accessed from any internet search engine when a question is written about the methods of anesthesia that can be applied during C/S. This information may have positive or negative effects on the patient, as well as include uncontrolled, unsupervised comments, articles and images. Our aim is primarily to evaluate whether our patients are exchanging information via social media or the internet and the effects of these shares on their concerns

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, who speaks and writes Turkish

Exclusion Criteria:

* psychiatric illness

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — caesarian section patients will be include
Study Population: caesarian section ASA I-II, who speaks and writes Turkish patients
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
social media effect on the anesthesia choice | were performed before the operation when the patient hospitalized.
  the effect of the uncontrolled disinformation on the patients decision of the anesthesia
social media and patient anxiety about anesthesia and surgery | before the operation when the patient hospitalized.
  anxiety will be measured

CONTACTS AND LOCATIONS:
Overall Officials: namık nebi ozcan, Study Chair — Ankara City Hospital Bilkent
Locations (2):
- Turkey (Türkiye) (2):
  - Aygün Güler, Ankara, Type A Choice Below ...
  - Ankara City Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asiodu IV, Waters CM, Dailey DE, Lee KA, Lyndon A. Breastfeeding and use of social media among first-time African American mothers. J Obstet Gynecol Neonatal Nurs. 2015 Mar-Apr;44(2):268-78. doi: 10.1111/1552-6909.12552. Epub 2015 Feb 24. PMID 25712127
- [Background] Gleeson DM, Craswell A, Jones CM. Women's use of social networking sites related to childbearing: An integrative review. Women Birth. 2019 Aug;32(4):294-302. doi: 10.1016/j.wombi.2018.10.010. Epub 2018 Dec 31. PMID 30606628
- [Background] Holtz B, Smock A, Reyes-Gastelum D. Connected Motherhood: Social Support for Moms and Moms-to-Be on Facebook. Telemed J E Health. 2015 May;21(5):415-21. doi: 10.1089/tmj.2014.0118. Epub 2015 Feb 9. PMID 25665177
- [Background] Pretorius K, Johnson KE, Rew L. An Integrative Review: Understanding Parental Use of Social Media to Influence Infant and Child Health. Matern Child Health J. 2019 Oct;23(10):1360-1370. doi: 10.1007/s10995-019-02781-w. PMID 31222601
- [Background] Barello S, Triberti S, Graffigna G, Libreri C, Serino S, Hibbard J, Riva G. eHealth for Patient Engagement: A Systematic Review. Front Psychol. 2016 Jan 8;6:2013. doi: 10.3389/fpsyg.2015.02013. eCollection 2015. PMID 26779108
- [Background] Field T. Prenatal anxiety effects: A review. Infant Behav Dev. 2017 Nov;49:120-128. doi: 10.1016/j.infbeh.2017.08.008. Epub 2017 Sep 5. PMID 28886563
- [Background] Perkin MR, Bland JM, Peacock JL, Anderson HR. The effect of anxiety and depression during pregnancy on obstetric complications. Br J Obstet Gynaecol. 1993 Jul;100(7):629-34. doi: 10.1111/j.1471-0528.1993.tb14228.x. PMID 8369244
- [Background] Che YJ, Gao YL, Jing J, Kuang Y, Zhang M. Effects of an Informational Video About Anesthesia on Pre- and Post-Elective Cesarean Section Anxiety and Recovery: A Randomized Controlled Trial. Med Sci Monit. 2020 Apr 8;26:e920428. doi: 10.12659/MSM.920428. PMID 32265432